CLINICAL TRIAL: NCT00074035
Title: A Phase II Trial Of Intravenous Pentostatin For The Treatment Of Patients With Refractory Chronic Graft-Versus-Host Disease
Brief Title: Pentostatin in Treating Patients With Refractory Chronic Graft-Versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CALGB-100101; U10CA031946 (NIH); CDR0000341678 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Pentostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pentostatin (Experimental): treatment of pts with refractory graft vs host disease
  Interventions: Drug: pentostatin

INTERVENTIONS:
Drug: pentostatin — 4 mg/sq m IV infusion over 20-30 min q 2 weeks

SUMMARY:
RATIONALE: Pentostatin may be effective in treating chronic graft-versus-host disease by stopping the immune system from rejecting donor stem cells or donor white blood cells.

PURPOSE: This phase II trial is studying how well pentostatin works in treating patients with chronic graft-versus-host disease that is refractory (not responsive) to treatment with steroids.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with refractory chronic graft-versus-host disease treated with pentostatin.

Secondary

* Determine the time to next immunosuppressive agent (i.e., the time to progression from best response) in patients treated with this drug.
* Determine the toxicity of this drug in these patients.
* Determine the infection rate in patients treated with this drug.
* Determine the pharmacokinetics of this drug in these patients.
* Determine the changes in lymphocyte populations in patients treated with this drug.
* Determine the survival of patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive pentostatin IV over 20-30 minutes on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients who achieve a complete response after 6 courses receive 4 additional courses. Patients who achieve a partial response, minor response, or stable disease after 6 courses may receive up to 6 additional courses.

Patients are followed every 4 weeks for 1 year, every 3 months for 2 years, and then annually for 5 years.

PROJECTED ACCRUAL: Approximately 37 patients will be accrued for this study.

ELIGIBILITY:
1. Histologic documentation of chronic GvHD following allogeneic HCT or donor lymphocyte infusion.
2. Patients may have progressive, quiescent, or de novo onset chronic GvHD.
3. Patients with extensive stage chronic GvHD requiring systemic immunosuppressive therapy are eligible. Patients with limited stage disease are excluded. Extensive stage is defined according to Seattle criteria (9) as either:

   * Generalized skin involvement or
   * Limited skin involvement or hepatic involvement with any one of the following:

     * Liver histology showing chronic progressive hepatitis, bridging necrosis or cirrhosis
     * Eye involvement (Schirmer's test with < 5 mm wetting)
     * Involvement of minor salivary glands or oral mucosa
     * Involvement of any other organ
4. Patients must have failed treatment with, or experience progression after, prior corticosteroids for extensive stage chronic GvHD, as defined below.

   4.1 Patients will be considered to have failed corticosteroids if they have any one of the following criteria:
   * Progressive disease or less than a minor response in any organ system despite 2 weeks on corticosteroid treatment at least 1 mg/kg methylprednisolone or equivalent.
   * Failure to achieve at least a minor response after at least 4 weeks of treatment with a dose of ≥ 0.5 mg/kg methylprednisolone or equivalent.
   * Achievement of less than a partial response at 8 weeks of corticosteroid treatment despite use of a dose ≥ 0.5 mg/kg methylprednisolone or equivalent.
   * Requirement of ≥ 0.5 mg/kg methylprednisolone or equivalent to maintain a partial response or better at 12 weeks of corticosteroid treatment.
   * Requirement of > 10 mg/kg methylprednisolone or equivalent to maintain a partial response or better at 18 weeks of corticosteroid treatment.

   4.2 Patients with progression of extensive stage chronic GvHD after a prior history of treatment with at least 18 weeks of corticosteroids, now requiring the reintroduction of corticosteroids (> 10 mg/day methylprednisolone or equivalent) or an additional agent (including photopheresis, PUVA) for treatment.
5. Patients with established chronic GvHD not improving or progressing on other immunosuppressive agents are also eligible if steroid refractoriness has been established previously.
6. Age ≥ 18 years
7. Performance Status 0-3
8. Patients on mechanical ventilation are excluded.
9. No active infection. Patients with active infection requiring antibiotic therapy are not eligible until infection is controlled.
10. No HIV infection. Patients with HIV infection are excluded because of safety concerns in this patient population.
11. Non-pregnant and non-nursing. Women and men of reproductive potential should agree to use an appropriate method of birth control throughout their participation in this study due to the teratogenic potential of the therapy utilized in this trial (although it is unlikely that successful pregnancy will occur in patients with chronic GvHD). Appropriate methods of birth control include oral contraceptives, implantable hormonal contraceptives (Norplant®), or double barrier method (diaphragm plus condom).
12. Required Initial Laboratory Values:

    * Calc. Creatinine Clearance ≥ 30 mL/min/1.73 m^2
    * ANC > 1000/μL
    * Platelets > 50,000/μL without transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-12 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2014-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif S. Farag, MD, PhD, Study Chair — Ohio State University
Locations (16):
- United States (16):
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2003 and March 2008, 39 participants were recruited to this study.
Pre-assignment Details: 1 participant cancelled prior to receiving treatment and is excluded from all analyses.
Groups:
- Pentostatin: pentostatin: 4 mg/m^2 IV infusion over 20-30 min q 2 weeks
Period: Overall Study
Arm/Group | Pentostatin
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 1 participant cancelled prior to receiving treatment and is excluded from all analyses.
Arm/Group | Pentostatin
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 48 [28 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 30
  More than one race | 1
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: count of participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Percentage of participants who had a complete or partial response defined by the Hopkins scoring system.
  A complete response is defined as the disappearance of signs and symptoms of chronic GVHD in all involved systems that is sustained for at lest 4 weeks. A partial response is an improvement by 2 or more points in at least one system score, which is sustained for at least 4 weeks, with no signs of worsening in others.
Time Frame: 3 months
Population: 3 patients died before the 3 month evaluation and were not evaluated for the primary endpoint
Measure: Number; unit: percentage of participants
Arm/Group | Pentostatin
Number analyzed (Participants) | 35
percentage of participants | 20

2. Secondary Outcome: Grade 3 or Higher Non-hematologic Adverse Events
Description: Number of participants experiencing a grade 3, 4 or 5 clinically significant non-hematologic adverse events, at least possibly related to treatment.
Time Frame: Duration of treatment (up to 5 years)
Measure: Number; unit: count of participants
Arm/Group | Pentostatin
Number analyzed (Participants) | 38
count of participants
  Fatigue | 3
  Renal failure | 4
  Anorexia | 2
  Infection | 10
  CNS hemmorrhage | 1
  Rash | 1
  Personality/behavioral | 1
  Pneumonitis | 1

3. Secondary Outcome: Overall Survival At 1 Year
Description: Percentage of patients who were alive at 1 year.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Pentostatin
Number analyzed (Participants) | 38
percentage of participants | 53

4. Secondary Outcome: Overall Survival At 2 Years
Description: Percentage of patients who were alive at 2 years.
Time Frame: 2 year
Measure: Number; unit: percentage of participants
Arm/Group | Pentostatin
Number analyzed (Participants) | 38
percentage of participants | 50

5. Other Pre Specified Outcome: Pharmacokinetics Association Between Exposure and Response At 3 Months
Description: The individual PK parameters will be derived by using a noncompartmental analysis of the plasma-concentration-time data
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: 34 participants were evaluable for adverse events
Arm/Group | Pentostatin
Serious Adverse Events (participants affected / at risk) | 14/34
Other Adverse Events (participants affected / at risk) | 30/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentostatin (N=34)
Hemoglobin decreased (Blood and lymphatic system disorders) | 11 (16)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Edema (Cardiac disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 4 (8)
Eye disorder (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (8)
Dry mouth (Gastrointestinal disorders) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (4)
Fever (General disorders) | 2 (2)
General symptom (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Localized edema (General disorders) | 2 (2)
Pain (General disorders) | 3 (3)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (4)
Immune system disorder (Immune system disorders) | 1 (2)
Catheter related infection (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 3 (4)
Opportunistic infection (Infections and infestations) | 1 (1)
Phlebitis infective (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 9 (15)
Alkaline phosphatase (Investigations) | 4 (8)
Alkaline phosphatase increased (Investigations) | 5 (7)
Aspartate aminotransferase increased (Investigations) | 11 (17)
Blood bilirubin increased (Investigations) | 7 (11)
Coagulopathy (Investigations) | 1 (1)
Creatinine increased (Investigations) | 8 (12)
Laboratory test abnormal (Investigations) | 4 (7)
Leukocyte count decreased (Investigations) | 7 (11)
Lymphocyte count decreased (Investigations) | 2 (3)
Neutrophil count decreased (Investigations) | 5 (5)
Platelet count decreased (Investigations) | 8 (11)
Serum cholesterol increased (Investigations) | 2 (2)
Weight loss (Investigations) | 2 (5)
Anorexia (Metabolism and nutrition disorders) | 4 (5)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 3 (6)
Blood glucose increased (Metabolism and nutrition disorders) | 7 (8)
Dehydration (Metabolism and nutrition disorders) | 5 (7)
Iron overload (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 7 (9)
Serum calcium decreased (Metabolism and nutrition disorders) | 7 (9)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 4 (7)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (3)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (4)
Serum potassium increased (Metabolism and nutrition disorders) | 3 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 6 (10)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (4)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (3)
Hypotension (Vascular disorders) | 3 (3)
Thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentostatin (N=34)
Hemoglobin decreased (Blood and lymphatic system disorders) | 15 (67)
Arrhythmia supraventricular (Cardiac disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Cardiac disorder (Cardiac disorders) | 3 (6)
Edema (Cardiac disorders) | 3 (13)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 4 (15)
Cushingoid (Endocrine disorders) | 1 (8)
Cataract (Eye disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 5 (19)
Extraocular muscle paresis (Eye disorders) | 1 (2)
Eye disorder (Eye disorders) | 2 (4)
Eye pain (Eye disorders) | 1 (2)
Glaucoma (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 3 (10)
Vision blurred (Eye disorders) | 4 (5)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 6 (20)
Diarrhea (Gastrointestinal disorders) | 9 (13)
Dry mouth (Gastrointestinal disorders) | 5 (10)
Dyspepsia (Gastrointestinal disorders) | 1 (4)
Dysphagia (Gastrointestinal disorders) | 3 (5)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 3 (7)
Esophageal stenosis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 3 (6)
Mucositis oral (Gastrointestinal disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 11 (22)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (9)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 3 (6)
Fatigue (General disorders) | 12 (33)
Fever (General disorders) | 3 (4)
Gait abnormal (General disorders) | 1 (1)
General symptom (General disorders) | 2 (3)
Ill-defined disorder (General disorders) | 1 (1)
Pain (General disorders) | 7 (23)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 2 (3)
Hypersensitivity (Immune system disorders) | 1 (1)
Immune system disorder (Immune system disorders) | 1 (5)
Bladder infection (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 2 (2)
Infection without neutropenia (Infections and infestations) | 4 (6)
Opportunistic infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Skin infection (Infections and infestations) | 1 (3)
Tooth infection (Infections and infestations) | 1 (2)
Upper respiratory infection (Infections and infestations) | 3 (7)
Ureteritis (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 20 (61)
Alkaline phosphatase (Investigations) | 7 (27)
Alkaline phosphatase increased (Investigations) | 7 (16)
Aspartate aminotransferase increased (Investigations) | 20 (72)
Bilirubin associated with graft versus host disease (GVHD) for BMT studies (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 6 (10)
Creatinine increased (Investigations) | 10 (23)
Gamma-glutamyltransferase increased (Investigations) | 1 (4)
INR increased (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 6 (27)
Leukocyte count decreased (Investigations) | 11 (28)
Lymphocyte count decreased (Investigations) | 5 (27)
Neutrophil count decreased (Investigations) | 7 (15)
Platelet count decreased (Investigations) | 15 (46)
Serum cholesterol increased (Investigations) | 4 (4)
Weight loss (Investigations) | 3 (6)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (6)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 3 (5)
Blood glucose increased (Metabolism and nutrition disorders) | 15 (71)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Iron overload (Metabolism and nutrition disorders) | 1 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 6 (11)
Serum calcium decreased (Metabolism and nutrition disorders) | 10 (13)
Serum calcium increased (Metabolism and nutrition disorders) | 2 (5)
Serum glucose decreased (Metabolism and nutrition disorders) | 4 (6)
Serum magnesium decreased (Metabolism and nutrition disorders) | 4 (8)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (4)
Serum phosphate decreased (Metabolism and nutrition disorders) | 3 (7)
Serum potassium decreased (Metabolism and nutrition disorders) | 5 (6)
Serum potassium increased (Metabolism and nutrition disorders) | 5 (13)
Serum sodium decreased (Metabolism and nutrition disorders) | 11 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint disorder (Musculoskeletal and connective tissue disorders) | 2 (5)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (6)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 5 (5)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (6)
Ataxia (Nervous system disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (3)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (5)
Neurological disorder NOS (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (11)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (12)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (7)
Insomnia (Psychiatric disorders) | 2 (3)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (4)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (3)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Reproductive tract disorder (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (6)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (5)
Rash desquamating (Skin and subcutaneous tissue disorders) | 11 (63)
Rash/desquamation associated with graft versus host disease (GVHD) for BMT studies (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 4 (20)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (2)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (8)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less